CLINICAL TRIAL: NCT02899533
Title: [18F]Fluoroestradiol (FES) PET/CT Imaging To Evaluate In Vivo ER In Patients With Pulmonary Arterial Hypertension (PAH)
Brief Title: [18F]FES PET/CT in PAH
Status: Terminated | Type: Observational
Why Stopped: The method did not help with assessing PAH and so the trial was terminated early.
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Other Study IDs: 824918
Record Dates: First submitted 2016-08-02; First posted 2016-09-14 (Estimated); Last update posted 2021-05-18 (Actual); Status verified 2021-05

CONDITIONS: Pulmonary Arterial Hypertension
Keywords: PAH; Pulmonary hypertension
MeSH Terms: conditions — Pulmonary Arterial Hypertension; Hypertension, Pulmonary | interventions — 16-fluoroestradiol

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- FES PET/CT scan: All subjects will receive an [18F]FES PET/CT scan.
  Interventions: Drug: [18F] FES

INTERVENTIONS:
Drug: [18F] FES — [18F] FES PET/CT scan, imaging tracer
  Other Names: [18F]fluoroestradiol

SUMMARY:
In this study positron emission tomography (PET/CT) imaging will be used to evaluate evaluation of estrogen receptor heterogeneity and functionality in Pulmonary Arterial Hypertension (PAH) using the investigational radiotracer [18F]fluoroestradiol (FES).

DETAILED DESCRIPTION:
This is a feasibility study of serial FES scanning in female patients with Pulmonary Arterial Hypertension (PAH) to determine whether patients have detectable changes in FES SUV following treatment with fulvestrant on the separate therapeutic protocol IRB# 824861 "Estrogen Receptor Antagonist in Patients with Pulmonary Arterial Hypertension (ERA PAH)". Subjects will undergo up to 2 [18F]FES PET/CT scans for this protocol. A baseline FES PET/CT will occur on Day 0 (-2 days) of the companion treatment trial prior to initiation of fulvestrant. The second FES PET/CT scan will occur on week 9 (63 ± 7 days) after initiation of fulvestrant. We will compare SUV values after fulvestrant to pre-treatment values.

ELIGIBILITY:
Inclusion Criteria:

* 1. Women who are post-menopausal, defined as one of the following

  1. > 50 years old and a) have not menstruated during the preceding 12 months per medical record review or self-report or b) have follicle-stimulating hormone levels > 40 IU/L at screening OR
  2. < 50 years and follicle-stimulating hormone levels > 40 IU/L at screening OR
  3. history of bilateral oophorectomy per medical record review or self-report.

  2. Diagnosis of Pulmonary Arterial Hypertension (PAH) per medical record review.

  3. Patients must be candidates to receive treatment on the companion therapeutic trial "Estrogen Receptor-α Inhibitor in Patients with Pulmonary Arterial Hypertension (ERA PAH)" (IRB# 824861 "ERA PAH")

  4. Participants must be informed of the investigational nature of this study and be willing to provide written informed consent and participate in this study in accordance with institutional and federal guidelines prior to study-specific procedures.

Exclusion Criteria:

* 1. Inability to tolerate imaging procedures in the opinion of an investigator or treating physician

  2. Serious or unstable medical or psychological conditions that, in the opinion of the investigator, would compromise the subject's safety or successful participation in the study.

  3. Ineligible for the therapeutic trial IRB# 824861 "ERA PAH" entitled "Estrogen Receptor Antagonist in Patients with Pulmonary Arterial Hypertension (ERA PAH)" (IRB# 824861 "ERA PAH")

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Females only
Study Population: Post-menopausal women with Pulmonary Arterial Hypertension
Sampling Method: Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2016-07; Primary Completion 2021-04-06 (Actual); Study Completion 2021-04-06 (Actual)

PRIMARY OUTCOMES:
Evaluate [18F]FES uptake in patients with Pulmonary Arterial Hypertension (PAH) before and after initiation of fulvestrant. | Change from Baseline [18F]FES uptake at 9 weeks.
  Patients will have a baseline FES PET/CT scan prior to the initiation of fulvestrant and a second FES PET/CT scan 9 weeks after the initiation of fulvestrant.

SECONDARY OUTCOMES:
FES uptake and change with treatment | baseline
  Evaluate baseline [18F]FES PET/CT uptake and change in uptake with fulvestrant in patients with PAH as a predictor of treatment response.
Change in FES compared to change in hematopoietic progenitor cells | 2 years
  Correlate change in [18F]FES uptake with changes in the number of circulating hematopoietic progenitor cells after the administration of fulvestrant in PAH.
Change in FES compared to change in hormone levels | 2 years
  Correlate change in [18F]FES uptake with changes in plasma hormone levels (pg/mL) after the administration of fulvestrant in PAH.
Change in FES compared to change in NT-proBNP | 2 years
  Correlate change in [18F]FES uptake with changes in NT-proBNP (pg/mL) after the administration of fulvestrant in PAH.
Change in FES compared to change in plasma biomarkers | 2 years
  Correlate change in [18F]FES uptake with changes in other plasma biomarkers (pg/mL) after the administration of fulvestrant in PAH.

CONTACTS AND LOCATIONS:
Overall Officials: David Mankoff, MD, PhD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania Hospital, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No